CLINICAL TRIAL: NCT01231360
Title: The Effect of Exercise Training on Skeletal Muscle Metabolism in Peripheral Artery Disease
Brief Title: The Effect of Exercise Training on Skeletal Muscle Metabolism in Peripheral Artery Disease (PAD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: American Heart Association (Other); Joslin Diabetes Center (Other)
Responsible Party: Principal Investigator, Reena Pande, MD, Instructor, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010p001107RP
Record Dates: First submitted 2010-10-28; First posted 2010-11-01 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Claudication
Keywords: claudication; peripheral artery disease; PAD
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Training (Active Comparator): Subjects randomized to exercise training will participate in a three-month treadmill exercise program in 1-hour training sessions three times per week as previously described. After a 5-minute warm-up period, exercise is initiated at a low workload of 2 mph at 0% grade. Subjects walk until moderate claudication severity develops, and then rest until the discomfort resolves, repeating until the total exercise period is completed. The intensity of the treadmill exercise is increased as tolerated by increasing walking speed by 0.5-1 mph and/or grade by 1-2%. Subjects are encouraged to continue the walking program at home for at least 30 minutes on two separate occasions each week.
  Interventions: Other: Exercise Training
- Normal routine (Active Comparator): Subjects randomized to the routine activity control group will be asked to keep a log of their daily activities and return to the Vascular Research Center at weeks 4, 8, and 12 at which time they will be asked to return their log and undergo repeat treadmill testing and complete the 6 minute walk test.
  Interventions: Other: Normal routine

INTERVENTIONS:
Other: Exercise Training — Subjects randomized to exercise training will participate in a three-month treadmill exercise program in 1-hour training sessions three times per week as previously described. After a 5-minute warm-up period, exercise is initiated at a low workload of 2 mph at 0% grade. Subjects walk until moderate claudication severity develops, and then rest until the discomfort resolves, repeating until the total exercise period is completed. The intensity of the treadmill exercise is increased as tolerated by increasing walking speed by 0.5-1 mph and/or grade by 1-2%. Subjects are encouraged to continue the walking program at home for at least 30 minutes on two separate occasions each week.
  Arms: Exercise Training
Other: Normal routine — Subjects randomized to the routine activity control group will be asked to keep a log of their daily activities and return to the Vascular Research Center at weeks 4, 8, and 12 at which time they will be asked to return their log and undergo repeat treadmill testing and complete the 6 minute walk test.
  Arms: Normal routine

SUMMARY:
Specific Aim 1: To test the hypothesis that subjects with PAD and intermittent claudication have altered expression of genes that regulate skeletal muscle metabolism.

Specific Aim 2: To test the hypothesis that exercise training improves calf skeletal muscle insulin resistance and genes that regulate skeletal muscle metabolic function in PAD patients with intermittent claudication.

ELIGIBILITY:
Inclusion Criteria:

* claudication symptoms
* ABI ≤ 0.9 in the symptomatic leg

Exclusion Criteria:

* diabetes
* impaired fasting glucose
* peripheral vascular intervention within the prior six months
* recent unstable angina
* myocardial infarction or stroke within the prior six months
* changes to their HMG-CoA reductase inhibitor (statin)within the past three months
* changes to pentoxifylline and/or cilostazol regimen within the past three months or anticipated to be necessary during the study
* are on Coumadin
* exercise limitations for reasons other than intermittent claudication (such as congestive heart failure, angina, chronic lung disease, or other disorders affecting the limb such as arthritis or neuropathy)
* rest pain or ulcers due to critical limb ischemia
* lower extremity amputation

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2010-10; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Expression of genes regulating skeletal muscle metabolism | 3 months

SECONDARY OUTCOMES:
Additional measures include skeletal muscle glucose uptake, measures of functional capacity, leg blood flow, and quality of life. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Reena Pande, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States